CLINICAL TRIAL: NCT06080464
Title: A Study of Clinician Satisfaction and Likelihood of Clinical Adoption of the VERABAND™
Brief Title: Clinician Satisfaction With the VERABAND™
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Arbor Medical Innovations, LLC (Unknown)
Responsible Party: Principal Investigator, Daniel Whibley, Assistant Professor, Physical Medicine and Rehabilitation, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00235976; 1U44NS122002 (NIH)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VERABAND information (Experimental): Consented patient participants will be given a VERABAND™ activity monitor during an initial clinic visit (baseline) and will then be tracked longitudinally after beginning a new pain treatment regime as part of their normal ongoing care. VERABAND™ activity data reports (including a summary broken down by week) will subsequently be provided to treating clinicians prior to each patient's follow-up clinic visit.
  The arm is all of the clinicians of the participants.
  Interventions: Other: VERABAND information

INTERVENTIONS:
Other: VERABAND information — The device, VERABAND™, activity data reports (including a summary broken down by week) will be provided to treating clinicians prior to each patient's follow-up clinic visit.

SUMMARY:
The VERABAND™ is a newly-developed, disposable, wearable activity monitor. The researchers will assess clinician satisfaction with the usability and likelihood of clinical adoption of the newly-developed, disposable, wearable activity monitor, across multiple clinical sites in the chronic low back pain (cLBP) population.

DETAILED DESCRIPTION:
A total of 340 cLBP patients (estimating n=300 completers) will be recruited and evaluated under an approved institutional review board (IRB) protocol by a total of 20 clinician participants distributed across multiple tertiary pain clinics. Consented patient participants will be given a VERABAND™ activity monitor during an initial clinic visit (baseline) and will then be tracked longitudinally after beginning a new pain treatment regime as part of their normal ongoing care. VERABAND™ activity data reports (including a summary broken down by week) will subsequently be provided to treating clinicians prior to each patient's follow-up clinic visit. The primary outcome will be clinician satisfaction with usability of the VERABAND™ system to support clinical cLBP management, regardless of the specific treatment(s) implemented or their analgesic effectiveness. Each clinician will complete a usability satisfaction survey at the end of each patient's episode of care, which allows for exploratory analyses to identify whether the VERABAND™ system is perceived to be more useful for specific patient phenotypes (e.g., those with higher levels of pain and/or disability or specific psychological characteristics).

ELIGIBILITY:
Any treating clinician at a recruiting tertiary pain clinic will be eligible to participate.

Patient participants must meet the following criteria:

Inclusion Criteria:

* Ambulatory
* Diagnosis of chronic low back pain (cLBP) according to the criteria of National Institute of Health (NIH) Task Force on Research Standards for cLBP
* Answering 'Yes' to the question: Does your low back pain interfere with your mobility?
* Starting any new non-surgical treatment or combination of treatments for cLBP as part of their normal ongoing care, including medications; physical therapy/exercise; integrated therapies (e.g., massage, acupuncture, yoga); cognitive- behavioral therapy; and/or interventional procedures (e.g., epidural steroid or facet joint injections)
* Willingness to wear a VERABAND™ continuously until their next clinic visit and return used devices in the mail.

Exclusion Criteria:

* Clinical findings suggesting the presence of ongoing systemic disease, including fever, weight loss, initiation of pain following major trauma, immunosuppression, intravenous drug use, recent bacterial infection, severe or persistent sensory or motor involvement of bowel, bladder, or lower extremity; or any condition that would greatly limit physical activity not due to pain.
* Inability to speak and write English.
* Visual or hearing difficulties that would preclude participation.
* Severe psychiatric disorders that in the opinion of the investigative team would interfere with participation in the study. This includes any active suicidal ideations or history of suicide attempts. Exclusions will be based on self-reported medical history or chart review and in accordance with Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria.
* Individuals receiving disability or compensation or involved in litigation.
* Scheduled surgery before follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Measure clinician satisfaction of the usability of the VERABAND™ using the System Usability Scale (SUS) | approximately 7 weeks
  The SUS is comprised of 10 statements: Each statement is accompanied by a five-point scale Likert response option. The SUS ranges from 10-50 and the higher scores indicate higher clinician satisfaction with usability.
Measure the likelihood of clinical adoption of the VERABAND™ using Item 1 of the System Usability Scale (SUS) | approximately 7 weeks
  The SUS item is a five-point scale Likert response ranging from 1-5. Higher scores indicate increase likelihood of clinical adoption of the VERABAND™

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Whibley, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No